CLINICAL TRIAL: NCT05211882
Title: Pilot Wait-list Randomized Controlled Trial of the ENABLE (Educate, Nurture, Advise, Before Life Ends) Intervention for Heart Failure (HF) Patients and Their Caregivers in Singapore
Brief Title: ENABLE (Educate, Nurture, Advise, Before Life Ends) Intervention for Heart Failure (HF) Patients and Their Caregivers in Singapore
Acronym: ENABLE-HF-SG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: Ministry of Health, Singapore (Other Government); National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ENABLE
Record Dates: First submitted 2022-01-02; First posted 2022-01-27 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure
Keywords: Palliative care; Patients; Caregivers; Distress thermometer (DT); Integrated Palliative Care Outcome Scale (IPOS); ENABLE (Educate, Nurture, Advise, Before Life Ends)
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate (Experimental): Participants in the intervention arm will start on the ENABLE program at point of randomization.
  Interventions: Other: Immediate ENABLE nurse coaching, on top of usual care
- Wait-list (delayed) (Experimental): Participants on wait-list will start ENABLE 6 months after randomization.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Immediate ENABLE nurse coaching, on top of usual care — Participants in the intervention arm will start on the ENABLE program at point of randomization
  Arms: Immediate
Other: Usual Care — Participants on wait-list will continue on usual care and only start ENABLE 6 months after randomization.
  Arms: Wait-list (delayed)

SUMMARY:
To pilot a culturally adapted version of ENABLE (6-month program) for Heart Failure (HF) patients and caregivers in the inpatient and outpatient setting in Singapore. The investigators aim to determine the feasibility of trial procedures and assess the acceptability and preliminary efficacy of ENABLE with a randomized wait-list controlled trial design.

DETAILED DESCRIPTION:
Palliative care improves quality of life (QOL) of patients and their caregivers. The ENABLE (Educate, Nurture, Advise Before Life Ends) intervention is a novel, nurse-led, structured, palliative care coaching program, developed in the United States for patients (and caregivers of patients) facing serious illnesses. It aims to empower patients and caregivers to manage their problems, prepare for the future, and has showed beneficial impact on patient and caregiver QOL.

The ENABLE coaching program is a potentially scalable means of delivering palliative care to a large population; as compared to the current local model of palliative care provision, which uses a resource intensive multidisciplinary care model that is not easily scalable and therefore unlikely to meet the growing needs of HF patients and caregivers locally. However, it is unclear if the ENABLE HF program will be culturally acceptable and efficacious in Singapore, in view of differing socio-cultural attitudes and expectations regarding healthcare and treatments, decision making and care planning.

Overall aim - To pilot a culturally adapted version of ENABLE (6-month program) for HF patients and caregivers in the inpatient and outpatient setting in Singapore.

Specific Aim 1 - Assessment of feasibility of trial procedures in the local HF population. Intervention arm participants will start on ENABLE after randomization, while wait-list participants will start on ENABLE after 6 months. The investigators will evaluate the percentage of eligible participant dyads who consent to participate and who are able to complete the ENABLE program. The investigators will also explore the percentage completion rate of patient and caregiver reported outcome measures.

- Hypothesis: The investigators hypothesize a-priori that 80% of eligible participant dyads will consent to participate and 80% of eligible participant dyads will be able to complete the ENABLE program.

Specific aim 2 - Assessment of acceptability of ENABLE. The investigators aim to study the acceptability of ENABLE to all patient-caregiver dyads. This will be done through evaluating the total scores of a satisfaction survey of all participants at the end of ENABLE.

- Hypothesis: The investigators hypothesize that at least 80% of all participants will find the ENABLE program acceptable.

Specific aim 3 - Assessment of the possible efficacy of ENABLE. The investigators will evaluate whether there is an efficacy signal that indicates ENABLE may improve patient QOL in the local HF context.

- Hypothesis: The investigators hypothesize that patient participants randomized to the intervention arm will have more improvement in their mean QOL scores after 6 months as compared to the wait-list control group.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for patients:

  1. 21 years or older.
  2. Able to communicate in English or Chinese.
  3. Have a diagnosis of HF (stage C or D) by the American College of Cardiology guidelines and be of New York Heart Association (NYHA) stage 2, 3 or 4 functional statuses.
  4. Have an expected prognosis of at least 6 months.
  5. Be on disease directed HF management.
  6. Have had a hospitalization event within 6 months prior to recruitment.
* Inclusion criteria for caregivers:

  1. 21 years or older.
  2. Able to communicate in English or Chinese.
  3. Is a direct family caregiver of the patient.

Exclusion Criteria:

* Exclusion criteria for patients:

  1. Patients who are unable to give informed consent
  2. Patients who are already known to a palliative care service.
* Exclusion criteria for caregivers:

  1. Caregivers who are unable to give informed consent.
  2. Caregivers who are domestic helpers.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2024-09-25 (Actual)

PRIMARY OUTCOMES:
Feasibility of trial procedures - percentage of patients and caregivers that are recruited, successfully randomized, and able to complete the ENABLE program | 6 months.
  The percentage of eligible participants that are able to be recruited, randomized and subsequently complete the ENABLE program will be calculated.
Acceptability of ENABLE program - through completion of the client satisfaction questionnaire (CSQ-4) | 6 months.
  The total score of the CSQ-4 will be calculated for each participant. For the assessment of acceptability, scores from participants from both intervention and wait-list control groups will be pooled, except for participants who drop out prior to starting ENABLE (for reasons unrelated to the ENABLE program). The minimum expected score per participant is 4, and the maximum expected score per participant is 16. A higher score indicates higher satisfaction.
The possible efficacy of the ENABLE program- through evaluating change in patient quality of life (QOL) at 6 months as compared to baseline (assessed using the Kansas City Cardiomyopathy Questionnaire - KCCQ) | 6 months.
  For the primary outcome of change in patient QOL, we will compare the change in the QOL from baseline to 6 months post randomization in the intervention group versus the change from baseline to 6 months post randomization in the control group. The difference between the intervention and wait-list control arm will be quantified as Cohen's d effect sizes to get an initial estimate of the efficacy of ENABLE. The minimum score on KCCQ is 0 and maximum possible score is 100. A higher score indicates a better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Shirlyn Neo, MBBS, MRCP (UK), MMed, FAMS, Principal Investigator — National Cancer Centre, Singapore
Locations (2):
- Singapore (2):
  - National Cancer Centre Singapore, Singapore
  - National Heart Centre Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No